CLINICAL TRIAL: NCT01323361
Title: Multi-centre Observational Pilot-study for Evaluation of Variation in CA-125 and Other Inflammatory Markers in the Perioperative Period of Laparoscopic Ventral Hernia Repair
Brief Title: CA125 Levels and Other Inflammatory Markers in Laparoscopic Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Jan Lambrecht, MD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010/3264-1 (REK); 2010/29472 (Other: Datainspectorate, Norway)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Hernia
Keywords: inflammation; laparoscopy; hernia; incisional; trauma
MeSH Terms: conditions — Hernia; Inflammation; Surgical Wound; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-immunosupressed (No Intervention): Normal population
  Interventions: Procedure: Laparoscopic ventral hernia repair

INTERVENTIONS:
Procedure: Laparoscopic ventral hernia repair — Patients operated with laparoscopic repair of ventral or incisional hernia

SUMMARY:
The study aims to show variation in CA-125 and other inflammatory markers assumed to be a response to trauma and peritoneal inflammation in the perioperative period of laparoscopic ventral hernia repair

DETAILED DESCRIPTION:
CA-125 and other inflammatory markers as body temperature, CRP, PCT, leucocytes and neutrophils measured pre- and post-operatively - correlated to trauma size i.e. area of dissection, mesh size, number of fixation points etc.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted for ventral or incisional hernia repair

Exclusion Criteria:

* Loss-of-domain
* ASA above III
* Liver failure
* Abnormal CA-125 prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Level of variation in inflammatory markers related to "trauma" impact | 6 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: jan r lambrecht, md, Study Director — Sykehuset Innlandet HF; ole m øyen, Dr. Med., Study Chair — Oslo University Hospital; erik trondsen, Dr. Med., Study Chair — Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo University Hospital, Rikshospitalet, Oslo, Akershus
  - Sykehuset Innlandet HF, Gjøvik, Oppland